## **Statistical Analysis Plan: Emotion-Diet Interactions in Pregnancy (PREDIP)**

NCT04430439

Date of document: 4/6/2020

## STATISTICAL DESIGN AND POWER ANALYSIS

Statistical Design: The statistical approach for each of the Specific Aims will be performed as follows:

<u>Aim 1a:</u> A cross-over study design will test the hypothesis that experimental exposure to a standardized psychosocial stress task will potentiate the postprandial metabolic response to the standardized meal. Each subject will represent her own control within the assigned meal group (low or high GI). A paired-samples t-test will be employed, using the model:  $E[Y_i] = \Delta AUC_i = (AUC_i)v1 - (AUC_i)v2$ 

where  $Y_i$  denotes the outcome measurement (change in AUC<sub>glu/ins</sub> or AUC<sub>FFA</sub>) on maternal i, and AUC<sub>i</sub> denotes the AUC for either metabolic outcome at a given laboratory visit; v1 or v2. As such, a test of the hypothesis that the above equations equals 0, represents a test that the effect of acute psychosocial stress exposure does not moderate the postprandial response to a standardized meal. A sensitivity analysis to estimate the difference in response by randomization sequence will ensure that the order of protocols does not confound the results.

<u>Aim 1b:</u> To explore the difference in the postprandial metabolic response following acute psychosocial stress exposure across meal types (low *vs* high GI), an independent sample t-test will be employed to compare the mean AUC<sub>glucose/insulin</sub> between the high GI and low GI groups.

<u>Aim 2:</u> To determine whether individual variation in biological stress reactivity (*i.e.*, AUC<sub>cortisol</sub> and AUC<sub>HRV</sub>) moderates the effect of acute psychosocial stress on the metabolic response to the standardized meal, a general linear model accounting for within subject correlation will be employed, according to the model:

$$E[Y_{ij}] = \beta_0 + \beta_1 STRESS_{ij} + \beta_2 REACT_{ij}$$

where  $Y_{ij}$  denotes the outcome change in the AUC<sub>i</sub> on maternal i, STRESS denotes the condition of exposure (stress vs no stress) to mother i on laboratory visit j, and REACT denotes stress reactivity, measured by AUC<sub>cortisol</sub> or AUC<sub>HRV</sub>. A test of  $H_0$ :  $\beta_1 = 0$  will test the hypothesis that mean AUC<sub>i</sub> (AUC<sub>gluc/ins</sub> and AUC<sub>FFA</sub>) differs by stress condition after adjustment for stress reactivity. An exchangeable correlation matrix will be assumed in the model.

**Power Analysis**: The primary outcome of the proposed research is the difference in the postprandial glucose/insulin response to a standardized meal (of either low or high GI) between the stress and non-stress conditions. Utilizing a cohort of 40 women in each meal group, it is estimated that the proposed study will have approximately 80% power to detect a 0.44 standard deviation difference in the mean within subject change in postprandial metabolic response (AUC<sub>glu/ins</sub> and AUC<sub>FFA</sub>), associated with the introduction of the stress paradigm.